CLINICAL TRIAL: NCT01590316
Title: SafeBoosC - Safeguarding the Brain of Our Smallest Children - an Investigator-initiated Randomised, Blinded, Multinational, Phase II Feasibility Clinical Trial on Near-infrared Spectroscopy Monitoring Combined With Defined Treatment Guidelines Versus Standard Monitoring and Treatment as Usual in Premature Infants
Brief Title: SafeBoosC - a Phase II Trial
Acronym: SafeBoosC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gorm Greisen (Other)
Responsible Party: Sponsor-Investigator, Gorm Greisen, Professor, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SB010512
Record Dates: First submitted 2012-05-01; First posted 2012-05-02 (Estimated); Last update posted 2018-04-12 (Actual); Status verified 2018-04

CONDITIONS: Brain Injuries; Infant, Premature
Keywords: Brain Injuries; Infant, Premature; Spectroscopy, Near-Infrared; Randomized Controlled Trial
MeSH Terms: conditions — Brain Injuries; Premature Birth

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cerebral NIRS oximetry + treatment guideline based on reading (Experimental)
  Interventions: Device: Cerebral NIRS oximetry
- Blinded cerebral NIRS oximetry (No Intervention)

INTERVENTIONS:
Device: Cerebral NIRS oximetry — Cerebral NIRS oximetry during the first 72 hours of life.
  Other Names: INVOS 5100C with adult SomaSensor (SAFB-SM) (Covidien); NIRO-200NX (Hamamatsy Photonics K.K.)
  Arms: Cerebral NIRS oximetry + treatment guideline based on reading

SUMMARY:
Background 25,000 infants are born extremely preterm every year in Europe. This group of infants carries a high risk of death and subsequent cerebral impairment for the infant, especially in the first 72 hours of life. Mortality is about 20%, and about 25% of survivors live with either cerebral palsy or low intelligence quotient. Preventative measures are keys to reducing mortality and morbidity in this population. There is evidence that the cerebral oxygenation time spent out of range (time with hypoxia or hyperoxia) is associated with poor outcome in infants. Near-infrared spectroscopy (NIRS) has been used to monitor tissue oxygenation since the mid-1980s, and quantification of oxygenation (rStO2) in a percentage from 0 to 100% has been possible for 10 years. From almost 400 preterm infants normal ranges of rStO2 has been determined to be from 55% to 85%. Still, there are no clinical trials and thus no solid evidence of the clinical utility of NIRS in preterm infants. Thus, research on the benefits and harms of cerebral monitoring using NIRS as a part of clinical management of premature infants is much needed.

Objectives The primary objective of the SafeBoosC trial is to examine if it is possible to stabilise the cerebral oxygenation of extremely preterm infants during the first 72 hours of life through the application of cerebral NIRS oximetry and implementation of an rStO2-specific clinical treatment guideline. We hypothesise that by using the specified treatment guideline to respond to cerebral monitoring readings outside the target range, we would reduce the burden of hypo- and hyperoxia and consequently reduce brain injury.

Trial design This is an investigator-initiated randomised, blinded, multinational, phase II feasibility clinical trial involving preterm infants from 12 European countries.

Inclusion criteria The inclusion criteria are: neonates born more than 12 weeks preterm (gestational age up to 27 weeks and 6 days); decision to conduct full life support; parental informed consent; and cerebral NIRS oximeter placed within 3 hours after birth.

Sample size With a 50% reduction of the area outside the normal range of oxygenation in %hours in the experimental group compared to the control group as the minimal clinically significant difference, a standard deviation of the area outside the normal range of 83.2 %hours, a type I error (alpha) of 5%, and a type II error of 0.05 (power of 95%) inclusion of 75 preterm infants in the experimental group and 75 preterm infants in the control group is required. The inclusion of twins are likely to decrease power, so it has been decided to increase sample size to 165 on a pragmatic basis of estimating intracluster correlation, control event rate, and incidence of twin births.

Intervention The premature infants will be randomised into one of two groups (experimental or control). Common is that both groups will have a cerebral oximeter monitoring device placed within three hours after birth. In the experimental group, the cerebral oxygenation reading is visible, and the infant will be treated accordingly using a defined treatment guideline. In the control group, the cerebral oxygenation reading is NOT visible, and the infant will be treated as usual.

Trial duration Monitoring by cerebral oximeter will be started as soon as possible and within 3 hours after birth and the intervention will last for 72 hours. Thereafter, each neonate will be followed up at term date (approximately three months after birth) and at 24 months after term date.

Outcome measures The primary outcome is the burden of hypo- and hyperoxia in %hours during the first 72 hours after birth. The secondary outcomes are brain activity on an amplitude-integrated electroencephalogram (aEEG), blood biomarkers (brain fatty acid binding protein (BFABP), neuroketal, and S100β), serious adverse reactions (SARs), severe brain injury, and all cause mortality at term date (approximately three months after birth). The exploratory outcomes are burden of hypoxia, burden of hyperoxia, neonatal morbidities, brain injury score on magnetic resonance imaging (MRI), number of therapies implemented during the intervention, physiological variables (mean blood pressure (BP), pulse oximeter oxygen saturation (SpO2), and partial pressure of carbon dioxide (pCO2)), and psychomotor impairment according to neurodevelopmental scales at 24 months after term date.

ELIGIBILITY:
Inclusion Criteria:

* Neonates born more than 12 weeks preterm (gestational age up to 27 weeks and 6 days).
* Decision to conduct full life support.
* Possibility to place cerebral NIRS oximeter within 3 hours after birth.
* Obtained parental signed written informed consent.

Exclusion Criteria:

* A clinical decision not to provide full life support.
* No possibility to place the cerebral NIRS oximeter within 3 hours after birth.
* Lack of parental signed written informed consent.

Max Age: 3 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 165 (Estimated)
Dates: Start 2012-06; Primary Completion 2013-12 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
The burden of hypo- and hyperoxia | 0-72 hours of life
  The burden of hypo- and hyperoxia in %hours during the first 72 hours after birth, i.e, the area outside the normal ranges of cerebral oxygenation of 55-85% as measured by NIRS.

SECONDARY OUTCOMES:
Brain activities on amplitude-integrated EEG as assessed by the interburst interval. | at 64 hours of life
Blood and urine biomarkers (brain fatty acid binding protein, neuroketal, and S100β). | at 6 and 64 hours of life
Brain injury assessed by cerebral ultrasound. | 1st, 7th, 14th, 35th day of life, and at term date
All-cause mortality | At term data and 24 months after term date
Serious adverse reactions | 0 - 7th day of life
  Serious adverse reactions (SAR): any adverse reaction that results in death, is life-threatening, requires prolongation of existing hospitalisation, results in persistent or significant disability or incapacity, or requires intervention to prevent permanent impairment or damage.

CONTACTS AND LOCATIONS:
Overall Officials: Gorm Greisen, MD, Principal Investigator — Rigshospitalet, Capitol Region of Denmark
Locations (1):
- Department of Neonatology, Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Archieving anonymized data at Danish Data Archieve

REFERENCES:
- [Derived] Riera J, Hyttel-Sorensen S, Bravo MC, Cabanas F, Lopez-Ortego P, Sanchez L, Ybarra M, Dempsey E, Greisen G, Austin T, Claris O, Fumagalli M, Gluud C, Lemmers P, Pichler G, Plomgaard AM, van Bel F, Wolf M, Pellicer A. The SafeBoosC phase II clinical trial: an analysis of the interventions related with the oximeter readings. Arch Dis Child Fetal Neonatal Ed. 2016 Jul;101(4):F333-8. doi: 10.1136/archdischild-2015-308829. Epub 2015 Dec 8. PMID 26645538
- [Derived] Hyttel-Sorensen S, Pellicer A, Alderliesten T, Austin T, van Bel F, Benders M, Claris O, Dempsey E, Franz AR, Fumagalli M, Gluud C, Grevstad B, Hagmann C, Lemmers P, van Oeveren W, Pichler G, Plomgaard AM, Riera J, Sanchez L, Winkel P, Wolf M, Greisen G. Cerebral near infrared spectroscopy oximetry in extremely preterm infants: phase II randomised clinical trial. BMJ. 2015 Jan 5;350:g7635. doi: 10.1136/bmj.g7635. PMID 25569128
- [Derived] Hyttel-Sorensen S, Austin T, van Bel F, Benders M, Claris O, Dempsey E, Fumagalli M, Greisen G, Grevstad B, Hagmann C, Hellstrom-Westas L, Lemmers P, Lindschou J, Naulaers G, van Oeveren W, Pellicer A, Pichler G, Roll C, Skoog M, Winkel P, Wolf M, Gluud C. A phase II randomized clinical trial on cerebral near-infrared spectroscopy plus a treatment guideline versus treatment as usual for extremely preterm infants during the first three days of life (SafeBoosC): study protocol for a randomized controlled trial. Trials. 2013 May 1;14:120. doi: 10.1186/1745-6215-14-120. PMID 23782447
- See also: Related Info — http://www.rigshospitalet.dk/menu/AFDELINGER/Juliane+Marie+Centret/Klinikker/Neonatalklinikken/Forskningihovedmenu/SafeboosC/